CLINICAL TRIAL: NCT04123041
Title: A Randomized, Open-Label, Cross-Over Study to Characterize the Nicotine Uptake and Subjective Effects With Use of JUUL Electronic Nicotine Delivery Systems With Multiple Flavors and Nicotine Concentrations, Usual Brand of Combustible Cigarettes, a Comparator E-Cigarette and Nicotine Gum in Adult Smokers
Brief Title: Characterize the Nicotine Uptake and Subjective Effects With Use of JUUL Electronic Nicotine Delivery Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juul Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PROT-00033
Record Dates: First submitted 2019-09-25; First posted 2019-10-10 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Electronic Cigarette Use; Tobacco Smoking
Keywords: Electronic Nicotine Delivery System; Combustible Cigarettes; Nicotine
MeSH Terms: conditions — Vaping; Tobacco Smoking

STUDY DESIGN:
Masking Description: The study is open label; however, subjects will be masked to the percentage of nicotine in JUUL products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Virginia Tobacco (Experimental): Subjects will use 5 products according to a randomized crossover assignment: JUUL 5% Virginia Tobacco ENDS, JUUL 3% Virginia Tobacco ENDS, Subject's UB combustible cigarette, Comparator e-cigarette, Nicorette White Ice Mint 4 mg nicotine polacrilex gum.
  Interventions: Other: JUUL ENDS, Combustible cigarette, comparator e-cigarette, Nicorette gum
- Mint (Experimental): Subjects will use 5 products according to a randomized crossover assignment: JUUL 5% Mint ENDS, JUUL 3% Mint ENDS, Subject's UB combustible cigarette, Comparator e-cigarette, Nicorette White Ice Mint 4 mg nicotine polacrilex gum.
  Interventions: Other: JUUL ENDS, Combustible cigarette, comparator e-cigarette, Nicorette gum
- Menthol (Experimental): Subjects will use 5 products according to a randomized crossover assignment: JUUL 5% Menthol ENDS, JUUL 3% Menthol ENDS, Subject's UB combustible cigarette, Comparator e-cigarette, Nicorette White Ice Mint 4 mg nicotine polacrilex gum.
  Interventions: Other: JUUL ENDS, Combustible cigarette, comparator e-cigarette, Nicorette gum
- Mango (Experimental): Subjects will use 5 products according to a randomized crossover assignment: JUUL 5% Mango ENDS, JUUL 3% Mango ENDS, Subject's UB combustible cigarette, Comparator e-cigarette, Nicorette White Ice Mint 4 mg nicotine polacrilex gum.
  Interventions: Other: JUUL ENDS, Combustible cigarette, comparator e-cigarette, Nicorette gum

INTERVENTIONS:
Other: JUUL ENDS, Combustible cigarette, comparator e-cigarette, Nicorette gum — JUUL ENDS and comparator e-cigarette will be used for 5 minutes ad libitum, one combustible cigarette will be used ad libitum, Nicorette gum will be used for 30 minutes ad libitum

SUMMARY:
The purpose of this study is to estimate nicotine uptake and assess subjective effects during ad libitum use sessions of 4 flavors of JUUL ENDS (also referred to as nicotine salt pod system; NSPS) products (i.e., Virginia Tobacco, Mint, Menthol and Mango) with 2 different nicotine concentrations. Subjective effects will also be assessed to gain an understanding of the user's experience during and after JUUL ENDS product use to evaluate the abuse liability of the products. The subject population will consist of healthy adult, male and female smokers, 21 to 65 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Provides voluntary consent to participate in this study documented on the signed informed consent form (ICF).
2. Adult, male or female smoker, 21 to 65 years of age, inclusive, at screening.
3. Has been a smoker for at least 12 months prior to screening. Brief periods of non-smoking (e.g., up to ~7 consecutive days due to illness, quit attempt (prior to 30 days of screening), participation in a study where smoking was prohibited) during the 12 months prior to screening will be permitted at the discretion of the Investigator.
4. Currently smokes an average of 10 or more king size or 100s manufactured combustible cigarettes per day (CPD; non-menthol or menthol), as reported at screening.
5. Has a positive urine cotinine (≥200 ng/mL) at screening.
6. Has an exhaled CO (carbon monoxide) >10 ppm at screening.
7. A female subject of childbearing potential must have been using 1 of the following forms of contraception, and agree to continue using it through completion of the study: hormonal (e.g., oral, vaginal ring, transdermal patch, implant, or injection) consistently for at least 3 months prior to check-in (Day -1); double barrier method (e.g., condom with spermicide, diaphragm with spermicide) at screening; intrauterine device for at least 3 months prior to check-in (Day -1); a partner who has been vasectomized for at least 6 months prior to check-in (Day -1); abstinence beginning at least 6 months prior to screening.
8. A female subject of non-childbearing potential must be postmenopausal with amenorrhea for at least 1 year prior to check-in (Day -1) and follicle-stimulating hormone (FSH) levels consistent with postmenopausal status or have undergone one of the following sterilization procedures at least 6 months prior to check-in (Day -1): hysteroscopic sterilization; bilateral tubal ligation or bilateral salpingectomy; hysterectomy; bilateral oophorectomy.
9. Is willing to comply with the requirements of the study, including a willingness to use the study products during the study.

Exclusion Criteria:

1. Has a history or presence of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or any other condition that, in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. Has a clinically significant abnormal finding on the physical examination, medical history, vital signs, ECG, or clinical laboratory results, in the opinion of an investigator.
3. Has a positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV).
4. Has had an acute illness (e.g., upper respiratory infection, viral infection) requiring treatment within 14 days prior to check-in (Day -1).
5. Has a fever (>100.5°F) at screening or check-in (Day -1).
6. Has a body mass index (BMI) >40.0 kg/m2 or <18.0 kg/m2 at screening.
7. Has a history of drug or alcohol abuse within 24 months of check-in (Day -1), as determined by an investigator.
8. Has or has a history of diabetes mellitus, asthma, or chronic obstructive pulmonary disease.
9. Has used prescription anti-diabetic medication and/or insulin therapy within 12 months prior to screening.
10. Has taken any medication for depression or asthma within 6 months prior to screening.
11. Has a systolic blood pressure <90 or >150 mmHg, diastolic blood pressure <40 or >95 mmHg, or heart rate <40 or >99 bpm at screening.
12. Has experienced an allergic reaction following previous e-cigarette use or with exposure to any primary components of the e-liquids (nicotine, flavor, benzoic acid, propylene glycol and glycerol).
13. Has an estimated creatinine clearance <70 mL/minute (using the Cockcroft-Gault equation) at screening.
14. Has a positive urine screen for alcohol or drugs of abuse at screening or check-in (Day -1).
15. If female, the subject is pregnant, has a positive pregnancy test at screening, is lactating, or intends to become pregnant during the time period from screening through the end of study.
16. Has used medications known to interact with cytochrome P450 (CYP) 2A6 (including, but not limited to, amiodarone, amlodipine, amobarbital, buprenorphine, clofibrate, clotrimazole, desipramine, disulfiram, entacapone, fenofibrate, isoniazid, ketoconazole, letrozole, methimazole, methoxsalen, metyrapone, miconazole, modafinil, orphenadrine, pentobarbital, phenobarbital, pilocarpine, primidone, propoxyphene, quinidine, rifampicin, rifampin, secobarbital, selegiline, sulconazole, tioconazole, tranylcypromine) within 14 days or 5 half-lives of the drug, whichever is longer, prior to check-in (Day -1).
17. Has used nicotine-containing products other than manufactured cigarettes (e.g., ENDS products, roll-your-own cigarettes, bidis, snuff, nicotine inhaler, pipe, cigar, chewing tobacco, nicotine patch, nicotine spray, nicotine lozenge, or nicotine gum) within 30 days prior to check-in (Day -1).
18. Has any prior history of JUUL product use prior to screening.
19. Has used any prescription smoking cessation treatments, including, but not limited to, varenicline (Chantix®) or bupropion (Zyban®) within 3 months prior to check-in (Day -1).
20. Negative response (i.e., unwilling to use or unable to tolerate; e.g., experiences AEs (adverse events) during the product trial that will prevent the subjects from continuing to use the study products as judged by the investigator) to any of the JUUL products at screening.
21. Is a self-reported puffer (i.e., adult smokers who draw smoke from the cigarette into the mouth and throat but do not inhale).
22. Is planning to quit smoking during the study or postponing (within 30 days of screening) a quit attempt in order to participate in the study.
23. Has donated plasma within 7 days prior to check-in.
24. Has donated blood or blood products (with the exception of plasma as noted above), had significant blood loss, or received whole blood or a blood product transfusion within 56 days prior to check-in (Day -1).
25. Has participated in a previous clinical study for an investigational drug, device, biologic, or tobacco product within 30 days prior to check-in (Day -1).
26. Is or has a first-degree relative (i.e., parent, sibling, child) who is a current employee of the study site.
27. Is or has a first-degree relative (i.e., parent, sibling, child) who is a current employee, shareholder, or is member of the board of directors of JUUL Labs, Inc.
28. In the opinion of the Investigator, the subject should not participate in this study.
29. Has previously taken part in, has been excluded or withdrawn from, or has completed this study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Nicotine uptake | 120 minutes
  Baseline-adjusted maximum plasma nicotine concentration [Cmax]
Product liking as measured by the Product-Liking Questionnaire | 60 minutes
  Maximum response to the Product-Liking Questionnaire (visual analog scale, range of "not at all" to "a great deal")

SECONDARY OUTCOMES:
Nicotine uptake | 120 minutes
  Time of the maximum post-baseline nicotine concentration
Nicotine uptake | 30 minutes
  Area under the nicotine concentration-time curve calculated using linear trapezoidal summation from time 0 to 30 minutes
Nicotine uptake | 60 minutes
  Area under the nicotine concentration-time curve calculated using linear trapezoidal summation from time 0 to 60 minutes
Nicotine uptake | 120 minutes
  Area under the nicotine concentration-time curve calculated using linear trapezoidal summation from time 0 to 120 minutes
The effects of nicotine exposure as measured by the Nicotine Withdrawal Questionnaire visual analog scale | 60 minutes
  Maximum response to the Nicotine Withdrawal Questionnaire (visual analog scale, range "not at all" to "extremely")
The effects of nicotine exposure as measured by the Product Direct Effects Questionnaire | 60 minutes
  Maximum response to the Product Direct Effects Questionnaire (visual analog scale, range "not at all" to "extremely")
Subjective product assessments as measured by the Modified Product Evaluation Scale | 60 minutes
  Subjective product assessments as measured by responses to the Modified Product Evaluation Scale (scale range of 1 [not at all] to 7 [extremely])
Likelihood of future product use as measured by the Future Intent to Use the Product Questionnaire | 60 minutes
  Maximum response to the Future Intent to Use the Product Questionnaire (visual analog scale range of "definitely would not" to "definitely would")
E-cigarette product use | 5 minutes
  Change in mass of e-cigarette pods/cartridges
Physiologic impact of product use as measured by blood pressure | 60 minutes
  Systolic and diastolic pressures
Physiologic impact of product use as measured by heart rate | 60 minutes
  Heart rate
Puff count during ad libitum (e-)cigarette use periods | 5 minutes
  Number of puffs taken during ad libitum use session
Safety and tolerability of short-term product use assessed by monitoring the incidence of product-use emergent adverse events | 14 days
  Safety and tolerability will be assessed by monitoring the incidence of product-use emergent adverse events.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Altasciences Clinical Kansas, Inc., Kansas City, Kansas
  - Central Kentucky Research Associates, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babb S, Malarcher A, Schauer G, Asman K, Jamal A. Quitting Smoking Among Adults - United States, 2000-2015. MMWR Morb Mortal Wkly Rep. 2017 Jan 6;65(52):1457-1464. doi: 10.15585/mmwr.mm6552a1. PMID 28056007
- [Background] D'Ruiz CD, Graff DW, Robinson E. Reductions in biomarkers of exposure, impacts on smoking urge and assessment of product use and tolerability in adult smokers following partial or complete substitution of cigarettes with electronic cigarettes. BMC Public Health. 2016 Jul 11;16:543. doi: 10.1186/s12889-016-3236-1. PMID 27401980
- [Background] Gottlieb S, Zeller M. A Nicotine-Focused Framework for Public Health. N Engl J Med. 2017 Sep 21;377(12):1111-1114. doi: 10.1056/NEJMp1707409. Epub 2017 Aug 16. No abstract available. PMID 28813211
- [Background] Hatsukami DK, Zhang Y, O'Connor RJ, Severson HH. Subjective responses to oral tobacco products: scale validation. Nicotine Tob Res. 2013 Jul;15(7):1259-64. doi: 10.1093/ntr/nts265. Epub 2012 Dec 13. PMID 23239843
- [Background] Jensen RP, Luo W, Pankow JF, Strongin RM, Peyton DH. Hidden formaldehyde in e-cigarette aerosols. N Engl J Med. 2015 Jan 22;372(4):392-4. doi: 10.1056/NEJMc1413069. No abstract available. PMID 25607446
- [Background] McNeill A [et al.] E-cigarettes: an evidence update. A report commissioned by Public Health England [Report]. - 2015.
- [Background] Polosa R, Morjaria J, Caponnetto P, Caruso M, Strano S, Battaglia E, Russo C. Effect of smoking abstinence and reduction in asthmatic smokers switching to electronic cigarettes: evidence for harm reversal. Int J Environ Res Public Health. 2014 May 8;11(5):4965-77. doi: 10.3390/ijerph110504965. PMID 24814944
- [Background] Tanner JA, Tyndale RF. Variation in CYP2A6 Activity and Personalized Medicine. J Pers Med. 2017 Dec 1;7(4):18. doi: 10.3390/jpm7040018. PMID 29194389
- [Background] USDHH US Department of Health and Human Services The Health Consequences of Smoking- 50 Years of Progress: A Report of the Surgeon General [Book] / ed. Health National Center for Chronic Disease Prevention and Health Promotion (US) Office on Smoking and. - 2014.
- [Background] Wang TW, Asman K, Gentzke AS, Cullen KA, Holder-Hayes E, Reyes-Guzman C, Jamal A, Neff L, King BA. Tobacco Product Use Among Adults - United States, 2017. MMWR Morb Mortal Wkly Rep. 2018 Nov 9;67(44):1225-1232. doi: 10.15585/mmwr.mm6744a2. PMID 30408019